CLINICAL TRIAL: NCT02618395
Title: Bioavailability Study of SPARC001 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUN-HBA-PK001
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: SPARC001A
- Treatment B (Experimental)
  Interventions: Drug: SPARC001B
- Treatment C (Experimental)
  Interventions: Drug: Reference001 - Hydrocodone

INTERVENTIONS:
Drug: SPARC001A
  Arms: Treatment A
Drug: SPARC001B
  Arms: Treatment B
Drug: Reference001 - Hydrocodone — Hydrocodone-acetaminophen
  Arms: Treatment C

SUMMARY:
Bioavailability study

DETAILED DESCRIPTION:
Bioavailability, safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Adult, male and female volunteers, 18 to 55 years of age
* Body mass index (BMI) ≥18 to ≤30 kg/m2 at screening
* Female subjects must have a negative serum pregnancy test
* Medically healthy on the basis of medical history and physical examination

Exclusion Criteria:

* Females who are pregnant, lactating, or likely to become pregnant during the study
* Life-time history and/or recent evidence of alcohol
* History of hypersensitivity to hydrocodone, acetaminophen or any component of the test and reference formulations
* Subjects with any condition in which an opioid is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
Maximum plasma hydrocodone and acetaminophen concentration (Cmax) | 17 days

SECONDARY OUTCOMES:
AUC extrapolated to infinity (AUC0 ∞) | 17 days
Time to Cmax (tmax) | 17 days
Elimination half-life (t½) | 17 days
Treatment emergent adverse event | 17 days